CLINICAL TRIAL: NCT07169799
Title: Evaluating the Impact of Cryotherapy Spray (Tru-Freeze) for the Eradication of Gastric Antral Vascular Ectasia (ICE-GAVE)
Brief Title: Impact of Cryotherapy Spray (Tru-Freeze) for the Eradication of Gastric Antral Vascular Ectasia (ICE-GAVE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Swathi Eluri, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-002286
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Gastric Antral Vascular Ectasia
MeSH Terms: conditions — Gastric Antral Vascular Ectasia

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm pre-post study with a 1:2 matched historical control cohort
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective arm: Spray Cryotherapy (Other): Subjects to receive baseline endoscopic confirmation/classification of GAVE, laboratory panels, and clinical indices. Once confirmed, subjects will undergo cryotherapy procedure schedule.
  Interventions: Other: trūFreeze® Spray Cryotherapy System (STERIS Endoscopy)

INTERVENTIONS:
Other: trūFreeze® Spray Cryotherapy System (STERIS Endoscopy) — This treatment consists of performing a diagnostic EGD to identify GAVE lesions. A catheter advances through the therapeutic channel to treat target areas with cryotherapy.
  Other Names: Procedure: EGD and truFreeze® spray-cryotherapy

SUMMARY:
The purpose of this study is to evaluate the impact of cryotherapy spray treatment for eradication of gastric antral vascular ectasia by measuring the change in hemoglobin levels and transfusion requirements in the first 6 months of cryotherapy treatment compared to the previous 6 months

ELIGIBILITY:
Inclusion Criteria

• Diagnosis of antral-predominant GAVE: Endoscopic confirmation of gastric-antral vascular ectasia affecting the antrum, without severe portal-hypertensive gastropathy. Sub-classify as nodular or non-nodular GAVE.

* Age: ≥ 18 years at the time of consent.
* Recent transfusion-dependent anemia

  * ≥ 1 packed-RBC transfusion for GAVE-related bleeding within the last 6 months to maintain hemoglobin (Hgb) > 8 g/dL (or > 7 g/dL if no coronary/vascular disease).
  * Standard-of-care transfusion thresholds:

    * If no coronary artery/vascular disease (CVD): transfuse 2 units when Hgb < 7 g/dL.
    * If CVD present: transfuse 2 units when Hgb < 8 g/dL.
    * After any transfusion, re-check Hgb within 1 week and repeat transfusion per the same criteria as needed.
* Documented transfusion history:

  o Medical records must show indication that each transfusion was for presumed GAVE-related bleeding.
* Treatment status:

  o Either treatment-naïve or ≤ 3 prior endoscopic ablation sessions for GAVE.
* Baseline data availability: Participant records must include endoscopic treatment dates, hemoglobin values, and transfusion data for 6 months prior to enrollment (extension up to 9 months permitted if data unavailable). Required elements:

  * total number of transfusions,
  * total number of prior endoscopic treatments, and calculated change in hemoglobin from baseline: Δ Hgb = Hgb(T-6 mo) - Hgb(T0) [extendable to Hgb(T-9 mo) if 6-month data are incomplete]
* Capacity to consent: Able and willing to provide written informed consent.

Exclusion Criteria

* Other gastrointestinal pathology

  o Active peptic-ulcer disease, inflammatory bowel disease, severe portal-hypertensive gastropathy, or untreated esophageal/gastric varices.
* Coagulopathy

  o Known bleeding disorder or acquired coagulopathy not attributable to GAVE.
* Severe comorbidity / high procedural risk

  * Advanced heart failure, severe renal impairment, or any condition classified ASA IV or V.
  * Estimated life-expectancy < 6 months.
  * Karnofsky performance status ≤ 40.
  * Deemed unfit for endoscopic procedures by the treating physician.
* Pregnancy / lactation:

  o Pregnant or breastfeeding, or planning pregnancy within 6 months of consent.
* Prior incompatible therapy

  o Previous cryoballoon ablation for GAVE.
* Ability to participate

  * Unable or unwilling to comply with the protocol or follow-up schedule.
  * Unable or unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-09-22 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical benefit of truFreeze® spray-cryotherapy in patients with gastric-antral vascular ectasia. | over 6 month period
  Changes in mean hemoglobin concentrations.
  Total number of packed-RCB units during a 6-month period after treatment and 6-months prior to treatment (retrospective review)

SECONDARY OUTCOMES:
Endoscopic success. | over 6 month period
  Endoscopic success (as assessed by independent endoscopic image review) measured safety of the cryotherapy procedure (adverse event tracking and assessments) change in means of patient's quality of life (measured by SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Eluri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials